CLINICAL TRIAL: NCT01344902
Title: An Open Dose-finding Study of Oral Applied Hexaminolevulinate (HAL) Imaging in Patients With Suspicion or High Risk of Neoplasia in the Colon
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to inadequate efficacy after 13 patients were evaluated.
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PC CO201/08
Record Dates: First submitted 2010-01-14; First posted 2011-04-29 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hexaminolevulinate (Experimental)
  Interventions: Drug: hexaminolevulinate HCl

INTERVENTIONS:
Drug: hexaminolevulinate HCl — 200mg hexaminolevulinate HCl capsule 6 hours before colonoscopy

SUMMARY:
The purpose of the study is to determine if it is possible to detect more pre-cancerous lesions in colon when using fluorescence technology.

DETAILED DESCRIPTION:
Carcinoma of the lower GI-tract is among the leading malignancies in the western world causing a substantial morbidity, mortality and consequently a large burden to the health care system in the diagnosis, treatment and follow-up of these patients.

The primary objectives of this study is to determine carcinoma- and adenoma lesion true detection rate of HAL fluorescence colonoscopy in patients with known or strong suspicion of neoplasia in the colon. The secondary objective and endpoints are to determine carcinoma- and adenoma lesion false detection rate of HAL fluorescence colonoscopy, to compare carcinoma- and adenoma lesion true detection rates and the false detection rates of fluorescence with standard colonoscopy and to characterize the safety profile of HAL fluorescence colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Female and Male subjects with known or strong suspicion iof adenoma or carcinoma of the colon after screening of follow-up colonoscopy
* Female and male patients with verified neoplastic lesions

Exclusion Criteria:

* Known or strong suspected porphyria
* Contraindications to colonoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine the carcinoma- and adenoma lesion true detection rate | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum München Pasing, Munich, Germany

REFERENCES:
- [Result] Mayinger B, Neumann F, Kastner C, Degitz K, Hahn EG, Schwab D. Early detection of premalignant conditions in the colon by fluorescence endoscopy using local sensitization with hexaminolevulinate. Endoscopy. 2008 Feb;40(2):106-9. doi: 10.1055/s-2007-967019. Epub 2008 Jan 16. PMID 18197583